CLINICAL TRIAL: NCT05449262
Title: Time Course Effects of Functional Resistance Training on Fitness and Quality of Life in Patients With Nonspecific Chronic Low-back Pain
Brief Title: Time Course Effects of Functional Resistance Training on Fitness and Quality of Life Chronic Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 01054 Hafiza Sana Asad
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Chronic Low-back Pain
Keywords: Pain; disability; strength; quality of life; functional resistance training
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- functional resistance training GROUP A (Experimental): Session of 45-60 min starting with Warm Up Exercise and stretching prior to therapy and cool-down and stretching after the training sessions
  Interventions: Other: functional resistance training GROUP A
- functional resistance training GROUP B (Experimental): Session of 45-60 min starting with Warm Up Exercise and stretching prior to therapy and cool-down and stretching after the training sessions
  Interventions: Other: functional resistance training GROUP B

INTERVENTIONS:
Other: functional resistance training GROUP A — Session of 45-60 min. Warm up prior to training Warm up 6-7 min of mild cardiovascular exercise followed by 3-4 min stretching
  Cool down post training A cool-down of 1 min of mild cardiovascular exercise followed by 4 min of stretching
  Arms: functional resistance training GROUP A
Other: functional resistance training GROUP B — Session of 45-60 min Warm up prior to training Warm up 6-7 min of mild cardiovascular exercise followed by 3-4 min stretching
  Cool down post training A cool-down of 1 min of mild cardiovascular exercise followed by 4 min of stretching
  Arms: functional resistance training GROUP B

SUMMARY:
Low back pain is categorized according to its duration as acute (<6 weeks), sub-acute (6 weeks - 12 weeks) and chronic (>12 weeks). Low back pain can be either specific or non-specific. Specific low back pain is because of specific spinal pathologies including; Malignancy, Infection, Osteoporotic Collapse, Fracture, Ankylosing Spondylitis or other inflammatory disorders and Cauda equina compression. About 19 in 20 cases of acute (sudden onset) low back pain are classed as 'non-specific' It is called 'non-specific' because it is usually not clear what is actually causing the pain or there is no specific problem or disease that can be identified as to the cause of the pain.Functional Resistance Training (FRT) involves multiplanar and multi joint resistance exercises that simulate movement patterns from everyday life and sport Functional training exercises tend to focus more on the coordination, technique, posture, and core engagement instead of on training loads.

DETAILED DESCRIPTION:
The lower back is also called the 'lumbosacral area' of the back. It is the part of the back between the bottom of the ribs and the top of the legs and is made up of the spine bones (vertebrae), discs, nerves, muscles and ligaments. Pain in this region is called low back pain. (1) Low back pain is categorized according to its duration as acute (<6 weeks), sub-acute (6 weeks - 12 weeks) and chronic (>12 weeks). About 19 in 20 cases of acute (sudden onset) low back pain are classed as 'non-specific' It is called 'non-specific' because it is usually not clear what is actually causing the pain or there is no specific problem or disease that can be identified as to the cause of the pain. It is said that cause may be a sprain (an over-stretch) of a ligament or muscle, minor problem with the disc between two vertebrae, or a minor problem with a small 'facet' joint between two vertebrae. It is not possible to identify these causes of the pain by tests. Therefore, it is usually impossible to say exactly where the pain is coming from, or exactly what is causing the pain. Sometimes a pain may develop immediately after lifting something heavy, or after an awkward twisting movement. Sometimes it can develop for no apparent reason. Some people just wake up one day with low back pain. Typically the pain is in one area of the lower back, but sometimes it spreads to one or both buttocks or thighs. Non-specific low back pain is 'mechanical' in the sense that it varies with posture or activity. In a small number of cases the pain persists for several months or longer. This is called chronic back pain. There is no test that can prove or confirm non-specific low back pain.

Non-specific low back pain is classed as chronic (persistent) if it lasts longer than six weeks. In some people it lasts for months, or even years. Symptoms may be constant. Non-specific low back pain affects people of all ages and is a leading contributor to disease burden worldwide.

The ACSM defines functional RT (FRT) as activities involving multiple muscle, joint, and planar activities that are closely related to activities of daily living, combining upper and lower body movements to use more of the body in each movement. Few studies have examined FRT, though initial results suggest that FRT is associated with higher caloric expenditure and similar muscular strength, endurance, and gains in flexibility compared with a TRT program.

Functional training is becoming increasingly popular within the fitness industry and has been considered to be a better alternative than traditional resistance training for improving various measures of muscular fitness including strength, endurance, coordination and balance. The verb form of the word "function" pertains to the performance of an action, work or activity. Thus, exercise training programs that are deemed to be "functional" should be designed to mimic tasks or activities that occur in a person's daily life to make training adaptations more transferable. Engaging in regular RT provides physical, physiological and psychological health benefits while providing additional bone health benefits. Although RT has greatly increased in popularity, other types of training aside from traditional RT (TRT) have yet to be examined. One such type of training, ''functional fitness,'' is defined by the ACSM as the use of strength training to improve balance and ease of living, and was in the top 10 fitness trends in 2018.

Functional Resistance Training (FRT) involves multiplanar and multi joint resistance exercises that simulate movement patterns from everyday life and sport Functional training exercises tend to focus more on the coordination, technique, posture, and core engagement instead of on training loads. The goal of FRT is not hypertrophy but to promote a potential motor problem in order to train dynamic stabilization. Appropriate functional exercises are those in which the lumbo-pelvic region remains aligned within the neutral zone by co-contraction of the muscles of the trunk, while other demands executed with the extremities are simultaneously and successfully fulfilled. This method of training usually includes: a) spinal stabilization exercises; b) balance and proprioceptive exercises; c) flexibility exercises; d) resistance training exercises.

Functional RT may be more feasible and accessible due to the minimal equipment needed and the flexibility to be performed in and out of a typical gym setting.

ELIGIBILITY:
Inclusion Criteria:

* Patient having low back pain as a primary complaint, without associated leg pain;
* Chronic pain (>= 3 months, >= 3 days/week)
* non- specific (soft tissue in origin)
* Patient having no history of formal exercise training.
* Learning proper technique under expert supervision
* Postural stability (static/dynamic)

Exclusion Criteria:

* Receiving concurrent treatments from another practitioner for LBP
* Congenital deformities of spine
* Neurological conditions (neuropathy, radiculopathy)
* Musculoskeletal conditions (fractures, atrophy, weakness)
* Cardiovascular, Nephrological conditions
* Contraindications to exercise
* Involved in workers' compensation claims;
* Medications other than analgesics and NSAIDS

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS)for pain: | 6 weeks
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain. it is scientifically evident that VAS is a reliable and valid scale in aged more than 18 years. In many studies it is proved that VAS is a reliable scale but for validity it showed moderate to strong correlation for pain measurement. assessment to be done at base line after 6 weeks and after detraining of 6 weeks
Visual analogue scale (VAS)for pain: | 12 weeks
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain. it is scientifically evident that VAS is a reliable and valid scale in aged more than 18 years. In many studies it is proved that VAS is a reliable scale but for validity it showed moderate to strong correlation for pain measurement. assessment to be done at base line after 12 weeks and after detraining of 12 weeks
Oswestry Disability Index (ODI) for disability: | 6 weeks
  Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. Thus, for every question not answered, the denominator is reduced by 5. The ODI can be used to assess both chronic and acute conditions of varying severity. It has high test-retest reliability and takes around 5min for a patient to complete. assessment to be done at base line after 6 weeks and after detraining of 6 weeks.
Oswestry Disability Index (ODI) for disability: | 12 weeks
  Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. Thus, for every question not answered, the denominator is reduced by 5. The ODI can be used to assess both chronic and acute conditions of varying severity. It has high test-retest reliability and takes around 5min for a patient to complete. assessment to be done at base line after 12 weeks and after detraining of 12 weeks.
SHORT FORM-36 for HRQOL | 6 weeks
  The Short form -36 covers eight different dimensions of HRQOL: physical functioning, social functioning, role limitations due to physical functioning (role functioning-physical), bodily gain, general mental health, role limitations due to emotional functioning (role functioning-emotional), vitality (energy and fatigue), and general health perception. Scores can be summed together from all domains with differing weightings to contribute to two summary scores, a physical component score and a mental component score. The study findings indicate that the SF-36 is a reliable and valid instrument for assessment of HRQoL in patients. assessment to be done at base line after 6 weeks and after detraining of 6 weeks.
SF-36 for HRQOL | 12 weeks
  The SF-36 covers eight different dimensions of HRQOL: physical functioning, social functioning, role limitations due to physical functioning (role functioning-physical), bodily gain, general mental health, role limitations due to emotional functioning (role functioning-emotional), vitality (energy and fatigue), and general health perception. Scores can be summed together from all domains with differing weightings to contribute to two summary scores, a physical component score and a mental component score. The study findings indicate that the SF-36 is a reliable and valid instrument for assessment of HRQoL in patients. assessment to be done at base line after 12 weeks and after detraining of 12 weeks.

SECONDARY OUTCOMES:
Physical fitness with flamingo test | 6 weeks
  The Flamingo Balance Test is total body balance test, and forms part of the Eurofit Testing Battery. This single leg balance test assesses the strength of the leg, pelvic, and trunk muscle as well as dynamic balance. purpose: To assess the ability to balance successfully on a single leg. assessment to be done at base line after 6 weeks and after detraining of 6 weeks.
Physical fitness with flamingo test | 12 weeks
  The Flamingo Balance Test is total body balance test, and forms part of the Testing Battery. This single leg balance test assesses the strength of the leg, pelvic, and trunk muscle as well as dynamic balance. purpose: To assess the ability to balance successfully on a single leg. assessment to be done at base line after 12 weeks and after detraining of 12 weeks
physical fitness with back endurance test: | 6 weeks
  The starting position is the patient/client adopting a half prone lying on a plinth with the superior edge of the iliac crest at the edge of the plinth and the arms crossed over the chest. The lower limbs are strategically stabilized with straps. The patient/client is asked to maintains the upper body in a horizontal position and the timer is started. The test ends if the patient/client can maintain the said position for 4 minutes or can no longer maintain the set position before 4 minutes elapses. The stop time is recorded. Assesment to be done at baseline after 6 weeks and detraining of 6 weeks.
physical fitness with back endurance test: | 12 weeks
  The starting position is the patient/client adopting a half prone lying on a plinth with the superior edge of the iliac crest at the edge of the plinth and the arms crossed over the chest. The lower limbs are strategically stabilized with straps. The patient/client is asked to maintains the upper body in a horizontal position and the timer is started. The test ends if the patient/client can maintain the said position for 4 minutes or can no longer maintain the set position before 4 minutes elapses. The stop time is recorded. Assessment to be done at baseline after 12 weeks and detraining of 12 weeks.
physical function with side bridge test | 6 weeks
  The trunk lateral endurance test, also called the side-bridge test, assesses muscular endurance of the lateral core muscles (i.e., transverse abdominis, obliques, quadratus lumborum, and erector spinae). This timed test involves static, isometric contractions of the lateral muscles on each side of the trunk that stabilize the spine. Assessment to be done at baseline after 6 weeks and detraining after 6 weeks.
physical function with side bridge test | 12 weeks
  The trunk lateral endurance test, also called the side-bridge test, assesses muscular endurance of the lateral core muscles (i.e., transverse abdominis, obliques, quadratus lumborum, and erector spinae). This timed test involves static, isometric contractions of the lateral muscles on each side of the trunk that stabilize the spine. Assessment to be done at baseline after 12 weeks and detraining after 12weeks.
physical function with abdominal curl-up test | 6 weeks
  The curl up test measures abdominal muscular strength and endurance of the abdominals and hip-flexors, important in back support and core stability. assessment to be done at baseline after 6 weeks and detraining after 6 weeks.
physical function with abdominal curl-up test | after 12 weeks
  The curl up test measures abdominal muscular strength and endurance of the abdominals and hip-flexors, important in back support and core stability. assessment to be done at baseline after 12 weeks and detraining after 12 weeks.
physical function with 60-s squat test: | 6 weeks
  To test lower body muscle endurance. Perform for the greatest possible number of repetitions in 1 min without carrying out assisted movements using other body segments assessment to be done at baseline after 6 weeks and detraining after 6 weeks.
physical function with 60-s squat test: | 12 weeks
  To test lower body muscle endurance. Perform for the greatest possible number of repetitions in 1 min without carrying out assisted movements using other body segments assessment to be done at baseline after 12 weeks and detraining after 12 weeks.
Biofeedback pressure unit | 6 weeks
  The unit consists of a combined gauge and inflation bulb connected to a pressure cell. Designed by physical therapists, the Stabilizer registers changing pressure in an air-filled pressure cell allowing body movements to be detected during exercise. The Pressure Biofeedback Unit is a reliable tool when utilized with a population of subjects that can perform the abdominal drawing-in test. assessment to be done at baseline after 6 weeks and detraining after 6 weeks
Biofeedback pressure unit | 12 weeks
  The unit consists of a combined gauge and inflation bulb connected to a pressure cell. Designed by physical therapists, the Stabilizer registers changing pressure in an air-filled pressure cell allowing body movements to be detected during exercise. The Pressure Biofeedback Unit is a reliable tool when utilized with a population of subjects that can perform the abdominal drawing-in test. Assessment to be done at baseline after 12 weeks and detraining after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No